CLINICAL TRIAL: NCT06039735
Title: Cardiac Toxicity and Prognostic Value of New Echocardiographic Indicators in the Treatment of Primary Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202306-015
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Echocardiography; Oncocardiology
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with previous untreated multiple myeloma: Patients diagnosed multiple myeloma by bone marrow cytology without previous chemotherapy and/or hematopoietic stem cell transplantation
  Interventions: Other: Chemotherapy and/or autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Other: Chemotherapy and/or autologous hematopoietic stem cell transplantation — Didn't interfere patients' treatment plan. Patients with chemotherapy (lenalidomide,bortezomib and dexamethasone) and/or autologous hematopoietic stem cell transplantation(ASCT) which is assessed by clinical doctors and only conventional treatments were used

SUMMARY:
Multiple myeloma (MM) is a malignant proliferative plasma cell disease, which accounts for approximately 10% and ranks secondly of hematological malignancies in many countries. It is more common in the middle-aged and elderly, and currently cannot be healed.

2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS) showed the quantitative definition table for cancer related cardiovascular toxicity (CTR-CVT) related to cancer treatment, which is crucial for understanding and balancing the absolute benefits of cancer treatment before and during treatment, including the implementation of primary preventive treatment, optimization of pre-existing cardiovascular diseases, dosage, frequency, and duration of tumor treatment, occurrence and severity of cardiovascular complications during treatment, as well as overall cumulative treatment received, time after treatment, and interactions with other cardiovascular diseases. However, current researches on adverse cardiac events in MM treatment mostly focus on follow-up of the therapeutic effects of certain drugs or comparison of short-term small sample ultrasound changes, but lacking systematic follow-up monitoring after treatment and the establishment of predictive models based on echocardiographic indicators.

This study aims to find the monitoring indicators in the early stage that are more sensitive in anti-tumor therapy for multiple myeloma patients by monitoring the changes in echocardiographic indicators after therapy. Based on the prognosis and adverse event occurrence in multiple myeloma patients, a predictive model for combining new ultrasound indicators with anti-tumor therapy for cardiac damage events and prognosis is established.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant proliferative plasma cell disease, which accounts for approximately 10% and ranks secondly of hematological malignancies in many countries. It is more common in the middle-aged and elderly, and currently cannot be healed.

2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS) showed the quantitative definition table for cancer related cardiovascular toxicity (CTR-CVT) related to cancer treatment, which is crucial for understanding and balancing the absolute benefits of cancer treatment before and during treatment, including the implementation of primary preventive treatment, optimization of pre-existing cardiovascular diseases, dosage, frequency, and duration of tumor treatment, occurrence and severity of cardiovascular complications during treatment, as well as overall cumulative treatment received, time after treatment, and interactions with other cardiovascular diseases. However, current researches on adverse cardiac events in MM treatment mostly focus on follow-up of the therapeutic effects of certain drugs or comparison of short-term small sample ultrasound changes, but lacking systematic follow-up monitoring after treatment and the establishment of predictive models based on echocardiographic indicators.

This study aims to find the monitoring indicators in the early stage that are more sensitive in anti-tumor therapy for multiple myeloma patients by monitoring the changes in echocardiographic indicators after therapy. The investigators plan to collect the clinical examination and echocardiographic images in the baseline and 3/6/12/36/60 months after treatment. After offline measurement, the investigators can get the changes of the structural and functional parameters, such as diameters, volumes, ejection fraction and strain of ventricle and atrium. Based on the prognosis and adverse event occurrence in multiple myeloma patients, a predictive model for combining new ultrasound indicators with anti-tumor therapy for cardiac damage events and prognosis is established.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old
2. Patients diagnosed multiple myeloma by bone marrow cytology
3. Trends to be hospitalized and treated by RVd induction therapy
4. Be able to complete at least 3-4 cycles treatment

Exclusion Criteria:

1. Simultaneously diagnosed myocardial amyloidosis or other systemic amyloidosis
2. Severe cardiovascular diseases such as myocardial infarction, heart failure, or previous surgery such as bypass grafting or valve replacement
3. Severe arrhythmia such as atrial fibrillation
4. Poor echocardiographic image quality

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 years old diagnosed multiple myeloma by bone marrow cytology without previous chemotherapy and/or hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Impaired systolic function of left ventricle or potential myocardial injury | During the study period and follow-up with 3/6/12/36/60 months
  LVEF≥50%, with a decrease of more than 15% in GLS compared with baseline, with/without an increase in diagnosed cardiac markers (cTnI/cTnT>99 percentile, BNP≥35pg/mL, NT-proBNP≥125pg/mL or significantly increased compared to baseline);Newly LVEF decreased more than 10% compared with baseline and is 40-49%; or newly LVEF decreased less than 10% and is 40-49%, accompanied by a decrease of more than 15% in GLS or an increase in one of the diagnosed cardiac markers including cTnI/cTnT, BNP and NT-proBNP mentioned above compared with baseline
Impaired systolic function of left ventricle | During the study period and follow-up with 3/6/12/36/60 months
  Newly diagnosed LVEF<40%

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
This study is a single center study and don't plan to share with others

REFERENCES:
- [Result] Cowan AJ, Green DJ, Kwok M, Lee S, Coffey DG, Holmberg LA, Tuazon S, Gopal AK, Libby EN. Diagnosis and Management of Multiple Myeloma: A Review. JAMA. 2022 Feb 1;327(5):464-477. doi: 10.1001/jama.2022.0003. PMID 35103762
- [Result] Erratum: 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS): Developed by the task force on cardio-oncology of the European Society of Cardiology (ESC). Eur Heart J Cardiovasc Imaging. 2023 May 31;24(6):e98. doi: 10.1093/ehjci/jead080. No abstract available. PMID 37076917
- [Result] Bishnoi R, Xie Z, Shah C, Bian J, Murthy HS, Wingard JR, Farhadfar N. Real-world experience of carfilzomib-associated cardiovascular adverse events: SEER-Medicare data set analysis. Cancer Med. 2021 Jan;10(1):70-78. doi: 10.1002/cam4.3568. Epub 2020 Nov 10. PMID 33169938
- [Result] Das A, Dasgupta S, Gong Y, Shah UA, Fradley MG, Cheng RK, Roy B, Guha A. Cardiotoxicity as an adverse effect of immunomodulatory drugs and proteasome inhibitors in multiple myeloma: A network meta-analysis of randomized clinical trials. Hematol Oncol. 2022 Apr;40(2):233-242. doi: 10.1002/hon.2959. Epub 2021 Dec 30. PMID 34940983
- [Result] Nakao S, Uchida M, Satoki A, Okamoto K, Uesawa Y, Shimizu T. Evaluation of Cardiac Adverse Events Associated with Carfilzomib Using a Japanese Real-World Database. Oncology. 2022;100(1):60-64. doi: 10.1159/000519687. Epub 2021 Oct 21. PMID 34673654
- [Result] Buck B, Kellett E, Addison D, Vallakati A. Carfilzomib-induced Cardiotoxicity: An Analysis of the FDA Adverse Event Reporting System (FAERS). J Saudi Heart Assoc. 2022 Aug 31;34(3):134-141. doi: 10.37616/2212-5043.1311. eCollection 2022. PMID 36127934
- [Result] Liu Z, Zhang L, Liu M, Wang F, Xiong Y, Tang Z, Li Q, Lu Q, Liang S, Niu T, Huang H. Myocardial Injury in Multiple Myeloma Patients With Preserved Left Ventricular Ejection Fraction: Noninvasive Left Ventricular Pressure-Strain Myocardial Work. Front Cardiovasc Med. 2022 Jan 20;8:782580. doi: 10.3389/fcvm.2021.782580. eCollection 2021. PMID 35127857